CLINICAL TRIAL: NCT06341751
Title: Psychological Treatment for Persistent Fatigue: a Feasibility Study
Brief Title: Psychological Treatment for Persistent Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry); The Swedish Research Council (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Elin Lindsäter, clinical psychologist, PhD, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00393-01
Record Dates: First submitted 2024-03-13; First posted 2024-04-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-07

CONDITIONS: Fatigue; Fatigue Syndrome, Chronic; Exhaustion; Syndrome
Keywords: Psychological treatment; Primary care; cognitive behavioral therapy; internet intervention; feasibility
MeSH Terms: conditions — Fatigue; Fatigue Syndrome, Chronic; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psychological treatment (Experimental): Blended treatment, i.e., both physical face-to-face sessions and internet-based asynchronous support. Treatment period is 4-6 months (6 months primary endpoint).
  Interventions: Behavioral: Psychological treatment for persistent fatigue

INTERVENTIONS:
Behavioral: Psychological treatment for persistent fatigue — The treatment consists of three main phases: 1) goal-setting; stabilizing sleep-wake patterns and even distribution of activities over the day (pacing). Attention-shifting and cognitive reappraisal 2. Gradual increase in physical activity followed by gradual increase in mental and social activity 3. Individual work to reach treatment goals.

SUMMARY:
This is a non-randomized pilot study to investigate the feasibility and acceptability of a transdiagnostic psychological intervention for primary care patients in Region Stockholm, Sweden, who suffer from persistent and disabling fatigue.

DETAILED DESCRIPTION:
Previous research indicates that fatigue is a transdiagnostic symptom dimension rather than a disorder-specific pathofysiology. Similar psychosocial mechanisms can contribute to the development and perpetuation of fatigue across medical conditions. Cognitive and behavioral interventions targeting these perpetuating mechanisms have been found effective in reducing fatigue severity and functional impairment in a range of different fatigue-dominated diagnostic groups. Based on these findings, the investigators have developed a transdiagnostic intervention for primary care patients who suffer from persistent fatigue, independent of primary diagnosis. The treatment is a psychological intervention based on cognitive and behavioral principles that is administered over a period of 4-6 months. Treatment material will be delivered via an online treatment platform and therapist support will be given both face-to-face and via written asynchronous text-messages in the online treatment platform.

This initial feasibility study is non-randomized, meaning that all included patients will recieve treatment.

The project could provide feasibility of a transdiagnostic treatment for primary care patients with severe and persistent fatigue across medical conditions. If the inclusion procedure, the data-collection procedure, and the treatment are feasible, a larger randomized clinical trial (RCT) studying treatment effect is called for. An adequately powered RCT could provide firm scientific support for a novel, scalable, and cost-effective way to deliver an evidence-based treatment for this large and currently under-treated patient group. This would have a desirable impact on patients, families, healthcare units, and society at large, given that fatigue is associated with substantial suffering and work-disability and that treatment guidelines are currently lacking.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-67
2. severe, functionally disabling fatigue as a central symptom for at least 3 months
3. The fatigue is not a direct effect of an active disease process motivating another treatment (e.g., hypo-/hyperthyroidism, anemia, cancer, dementia) or the effect of medication
4. regular access to a computer and to the Internet
5. ability to read and write in Swedish.

Exclusion Criteria:

1. substance abuse disorder in the past 6 months
2. Current or past psychosis or bipolar disorder
3. Primary psychiatric disorder of such severity that it merits evidence-based treatment (e.g., obsessive compulsive disorder, moderate to severe depression, post-traumatic stress disorder)
4. elevated risk for suicide
5. anorexia nervosa
6. BMI>40
7. Initiated or changed psychopharmacological medication (e.g., for depression or anxiety disorders) in the past month
8. ongoing chemotherapy
9. intellectual disability (e.g., severe autism) that affects ability to work with the treatment
10. self-harm
11. pregnancy
12. life circumstances that complicate or make treatment impossible (e.g., domestic violence or ongoing legal disputes)
13. ongoing psychological treatment and/or multimodal rehabilitation.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In the initial screening, patients are asked to respond to the following question:
  "What is your gender? (with gender, we mean gender-identity, that is - your self-representation of gender)"
  Response-alternatives:
  Male Female Non-binary Other alternative Not sure Prefer not to answer
Enrollment: 18 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Treatment adherence and completion | Post-treatment (6 months)
  Treatment adherence will be assessed by evaluating how many sessions (face-to-face and video-based) the patient received, how many modules of the internet-delivered material the patient accessed, and the amount of time the patient spent in the online treatment platform (data extracted from the platform).
  Further, number of drop-outs (i.e., patients who discontinued treatment before treatment completion) will be analyzed
Treatment credibility | Three weeks after treatment start
  Assessed using the Credibility/Expectancy Questionnaire (C-Scale). The C-Scale is a 5-item measure, scale range is 0 to 50 points with higher scores indicating higher treatment credibility.
Patient satisfaction | Post-treatment (6 months)
  Client Satisfaction Questionnaire (CSQ-8). Total scores range from 8 to 32, with higher scores indicating greater treatment satisfaction.
Working alliance | Week 3 and 15 of treatment
  Assessed using the Working Alliance Questionnaire (WAI - short version). Scale range is from 6 to 42 with higher scores indicating a better percieved working alliance.
Negative effects of treatment | Post-treatment (6 months)
  The Negative Effects of Treatment Questionnaire (NEQ-20). The self-report measure consists of three parts. First, respondents endorse specific items in case they have occurred or not during treatment, yes/no (dummy coded as a variable: 1/0). Second, the respondents rate how negatively the negative effect was on four-point Likert-scale, ranging from "Not at all" to "Extremely", 0-4 ("0" being minimum and "4" being maximum). Third, the respondents attribute the negative effect to "The treatment I received" (1) or "Other circumstances" (0) (dummy coded as a variable: 1/0).
Open-ended questions regarding treatment content and presentation | Post-treatment (6 months)
  Post-treatment, patients will be asked open-ended questions regarding their perception of the different components of the treatment, how much time they spent working with the treatment, and their thoughts about the usability of the digital platform.

SECONDARY OUTCOMES:
Feasibility of study inclusion procedures and data-collection | Data will be collected during the recruitment and inclusion phase of the study.
  The recruitment procedure will be evaluated by accessing data from ALMA (a fully automated clinical desicion-support in the medical journal). ALMA aggregates anonymous data regarding number of times the algorithm has been activated and the number of times it has resulted in a referral to the study platform where screening for study inclusion is completed. Of those who complete screening, we will assess the proportion of patients who are included or excluded in the study.
  Data-collection procedures will be assessed by evaluating data-attrition at the various measurement points.
Fatigue severity, primary self-rated symptom outcome | Assessed pre- and at post treatment (6 months), and every three weeks during the treatment phase.
  Fatigue severity (self-rated) using the Checklist Individual Strenghts- Fatigue severity subscale. The domain Fatigue severity contains 8 items scored on a 7-point Likert scale (range 8-56; higher scores=more severe fatigue). A score above 35 points on the CIS-F indicates severe fatigue.
Problems concentrating | Assessed pre- and at post treatment (6 months)
  Subscale in the Checklist Individual Strengths Questionnaire (CIS), 5 items. Scale range: 5 to 35 with higher scores representing more problems concentrating.
Reduced physical activity | Assessed pre- and at post treatment (6 months)
  Subscale in the Checklist Individual Strengths Questionnaire (CIS), 3 items. Scale range: 3 to 21 with higher scores representing less physical activity.
Reduced motivation | Assessed pre- and at post treatment (6 months)
  Subscale in the Checklist Individual Strengths Questionnaire (CIS), 4 items. Scale range: 4 to 28 with higher scores representing less motivation.
Depressive symptoms | Assessed pre- and at post treatment (6 months). The individual item assessing suicide risk will be administered every 3 weeks during the traetment phase.
  Patient Health Questionnaire-9 (PHQ-9). Scale range is from 0 to 27, higher scores representing more depressive symptoms Note: the suicide-item will be administered every three weeks during the treatment phase.
Somatic symptoms | Assessed pre- and at post treatment (6 months)
  Physical Health Questionnaire-15 (PHQ-15). Scale range is from 0 to 30, higher scores representing more somatic symptoms
General anxiety | Assessed pre- and at post treatment (6 months)
  The General Anxiety Questionnaire (GAD-7). Scale range is from 0 to 21, higher scores representing more anxiety.
Insomnia | Assessed pre- and at post treatment (6 months), and every three weeks during the treatment phase.
  The Insomnia Severity Inventory (ISI) 7 items. Scale range is from 0 to 28, higher scores representing higher insomnia severity.
  NOTE: an additional item will be added to assess hypersomnia.
Perceived Stress | Assessed pre- and at post treatment (6 months)
  The Perceived Stress Scale (PSS-10). Scale range is from 0 to 40, higher scores representing a higher level of perceived stress.
Burnout | Assessed pre- and at post treatment (6 months)
  The Shirom-Melamed Burnout Questionnaire (SMBQ-18). Scale range is from 0 to 6, higher scores representing a higher level of burnout.
Self-rated health | Assessed pre- and at post treatment (6 months)
  The Self-rated health questionnaire (SRH-5). A single item with 5 response-categories, 0 (very bad health); 4 (very good health)
Cognitive and behavioral responses to symptoms | Assessed pre- and at post treatment (6 months), and every three weeks during the treatment phase.
  Cognitive and Behavioral Responses to Symptoms Questionnaire (CBRQ), 18-items. The scale assesses six domains: Fear avoidance (3 items, scale range 0-12); Damage beliefs (3 items, scale range 0-12); Embarrassment avoidance (3 items, scale range 0-12); Symptom focusing (3 items, scale range 0-12); All-or-nothing behaviour (3 items, scale range 0-12); Resting behaviour (3 items, scale range 0-12).
General self-efficacy | Assessed pre- and at post treatment (6 months), and every three weeks during the treatment phase.
  The General self-efficacy scale (GSE), 10 items. Scale range is from 10 to 40, higher scores representing a higher level of self-efficacy.
Functional disability | Assessed pre- and at post treatment (6 months)
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), 12 items. Scoring from 0 (maximum functional disability) to 100 (no functional disability)
Work and Social Adjustment | Assessed pre- and at post treatment (6 months)
  the Work and Social Adjustment Scale (WSAS), 5 items. Scale range 0 to 40 with higher scores representing better work and social adjustment.

OTHER OUTCOMES:
Treatment fidelity | Continuously throughout the 6-month treatment phase
  Treatment fidelity will be assessed by audio recording all synchronous treatment sessions, of which a random selection will be assessed for fidelity using checklists that correspond to the central treatment components in each phase of the treatment.
Evaluation of participants' experience of treatment | Post-treatment completion (at 6 months)
  When all treatments have been completed in the study, semi-structured interviews will be conducted with up to 10 included patients and up to three therapists. These will tap deeper, qualitative information about perceptions of working with the treatment and the data-collection procedures. All interviews will be audio recorded and transcribed for thematic content analysis.
Acceptability, Appropriateness, and Feasibility from the perspective of the clinic | Assessed post-treatment completion (after 6 months)
  a survey based on the "Triple P Systems Implementation Outcomes: Acceptability, Appropriateness, and Feasibility of intervention measure" will be disseminated to healthcare staff at participating primary health care clinics, to which they respond anonymously.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Lindsäter, PhD, Principal Investigator — Region Stockholm and Karolinska Institutet
Locations (1):
- Gustavsberg University Primary Care Clinic, Stockholm, Stockholm County, Sweden